CLINICAL TRIAL: NCT01273324
Title: Prospective Clinical Study Using Radiostereometric Analysis (RSA) and DEXA to Evaluate Fixation and Wear of the Restoration ADM Acetabular System
Brief Title: Radiostereometric Analysis (RSA) and DEXA to Evaluate Fixation and Wear of the Restoration ADM Acetabular System
Status: Completed | Type: Observational
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Michael Dunbar, MD, PhD, Dalhousie University
Other Study IDs: CDHA-RS/2012-079
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADM: ADM Cup
  Interventions: Device: ADM Cup

INTERVENTIONS:
Device: ADM Cup — ADM Cup
  Other Names: Styrker ADM Acetabular Cup

SUMMARY:
The dual mobility design concept for acetabular liners, as is used in the Restoration ADM Acetabular System, has been applied in various implants since its introduction by Gilles Bousquet in France in 1976. Dual mobility cups have shown good clinical results and have been particularly lauded for low incidence of dislocations. However, the wear performance of this design concept has not been proven to date. As wear particles are a possible contributing factor in aseptic loosening, the assessment of wear and fixation is an important step in proving this implant design.

The proposed study will combine RSA and peri-prosthetic bone mineral density as well as outcome questionnaires to provide a complete in vivo evaluation of prosthesis fixation, polyethylene wear, and objective and subjective outcomes for the Restoration ADM Acetabular System.

DETAILED DESCRIPTION:
Question 1: a) Do the implant components of the Restoration ADM Acetabular System achieve adequate fixation to the underlying bone? Null Hypothesis: There is no significant increase in micromotion of the implant components after 1 year indicating adequate long-term fixation at the implant - bone interface. Alternative Hypothesis: There is a significant increase in micromotion of of the implant components after 1 year indicating inadequate fixation at the implant - bone interface. b) What are the migration patterns (translations and rotations) of the Restoration ADM Acetabular System components during the first three years postoperatively? c) For what proportion of implants does migration continue to increase during the three year follow-up? d) Are inducible displacements, measured during weight-bearing follow-up exams, consistent over time and do they indicate that adequate fixation has been achieved? e) Are there significant differences in migration patterns (translations and rotations) between the Restoration ADM Acetabular System components and other implants previously studied with RSA and reported in the literature? Question 2: a) How much does the femoral head wear into the polyethylene liner?b)How much backside wear occurs on the polyethylene liner? c)How does the total wear compare to that with other implants previously reported in the literature? Question 3: Does the polyethylene liner demonstrate mobile bearing properties? Question 4: a) Are there changes over time in bone mineral density of peri-prosthetic bone with the Restoration ADM Acetabular System components? b) Where do changes in bone mineral density occur? Question 5: Does total hip arthroplasty using the Restoration ADM Acetabular System result in significant improvement in health status and functional outcome?

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic osteoarthritis of the hip indicating primary total hip arthroplasty
2. Between the ages of 21 and 80 inclusive
3. Patients willing and able to comply with follow-up requirements and self-evaluations
4. Ability to give informed consent

Exclusion Criteria:

1. Inflammatory arthritis
2. BMI >40
3. Post-traumatic arthritis of the hip
4. Prior arthroplasty with the affected hip
5. Hip dysplasia
6. Active or prior infection
7. Medical condition precluding major surgery
8. Severe osteoporosis or osteopenia

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoarthritis of the hip
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
RSA migration | 3 years

SECONDARY OUTCOMES:
RSA wear | 3 years
Questionnaires | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunbar, MD, FRCSC, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada